CLINICAL TRIAL: NCT01843517
Title: Endogenous Pain Facilitation and Inhibition in Postpartum Women
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00022603
Record Dates: First submitted 2013-04-25; First posted 2013-04-30 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Pain Inhibition and Facilitation in Post Partum Women
Keywords: Pain; Facilitation; Inhibition; Oxytocin; Postpartum
MeSH Terms: conditions — Pain; Inhibition, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- endogenous pain facilitation: Pain facilitation is studied by a simple test of applying over the counter capsaicin cream to the skin for only 30 min, then removing it and heating the skin to a non-noxious temperature.
- endogenous pain inhibition: Pain inhibition is studied by a simple test of mild pain on one area of the body reducing response to a pain stimulus in another area.

SUMMARY:
This study seeks to further understand these three observations - (1) that the time period surrounding childbirth accelerates recovery from pain after injury (2) that this likely reflects dampened facilitating mechanisms and exaggerated inhibitory mechanisms, and (3) that stress may interfere with this protection. In this study the investigators will compare women within 2 weeks of delivery to age matched controls and anticipate that pain inhibition is increased after delivery, pain facilitation is decreased, and that there is a relationship between these pain responses and the degree of pre-existing stress.

DETAILED DESCRIPTION:
Nearly half of the world's population experiences labor and delivery processes which are associated with microscopic or gross tissue injury to the mother. Since this experience is widespread and occurs relatively early in life, the psychosocial, medical, and financial consequences of chronic pain following childbirth could be enormous. Surprisingly, previous studies with long term follow up of new mothers have included pain as a secondary measure and / or have focused on prevalence of pain without determining whether pain predated delivery or even pregnancy itself. The investigators recently performed a long term follow up study of over 1,200 women, and noted that pain which began during the childbirth itself was surprisingly rare in comparison to other physical injuries. Additionally, two central factors hypothesized to confer risk of chronic pain after other injuries including surgery, pre-dating chronic pain and degree of tissue and nerve injury, contributed minimally to the acute and sub-acute pain after childbirth. These two observations, low incidence of chronic pain and minimal effect of degree of tissue injury and history of chronic pain on sub-acute pain, point towards a potential protective effect of pregnancy or delivery on the response to physical injury.

ELIGIBILITY:
Inclusion Criteria:

* female
* 10-14 days postpartum, term vaginal delivery
* breastfeeding (postpartum women)
* health non-pregnant female (nulliparous or at least 1 year beyond delivery)

Exclusion Criteria:

* Allergy to chili peppers
* pregnant
* pain medication (narcotic or non-narcotic) within 4 hours of study visit Average pain in the 24 hours preceding the study visit >3. Postpartum women that score >13 on the Edinburgh Postnatal Depression Scale

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women 10-14 days postpartum following term vaginal delivery, who are breast feeding and age- and race- matched healthy, nonpregnant women, either nulliparous or at least 1 year beyond delivery.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Area of hyperalgesia will be the primary outcome measure | 40 minutes post capsaicin application
  Hyperalgesia and allodynia on the skin of the forearm will be established by heating the forearm with a 4 cm2 Peltier controlled thermode (TSA®) to 45 degrees Celsius for 5 minutes. The investigators will then apply topical capsaicin (0.075% cream, Bioglan Pharmaceuticals) under an occlusive dressing at the same site as the thermal probe for 30 minutes. 40 minutes after removal of the capsaicin cream the site will be heated to 40 degrees Celsius for 5 minutes (rekindling) following the end of capsaicin application. The investigators will test skin sensations with the filament and cotton wisp after this heating.
Percent reduction in degree of pain to the 49 degrees Celsius stimulus during the time the foot is immersed in the cold water | 15 minutes
  Conditioned pain modulation will be induced by placing a foot in a container of circulating water maintained at 10 degrees Celsius for 90 seconds. Thirty seconds after the foot is placed into container of circulating water, the stimulus response to heat on the contralateral forearm will be measured using a 49 degrees Celsius stimulus for 5 seconds. The foot will then be withdrawn and warmed with warm blankets. The stimulus response to heat stimuli on the arm will be measured 5 and 15 min thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: James C. Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Pan PH, Tonidandel AM, Aschenbrenner CA, Houle TT, Harris LC, Eisenach JC. Predicting acute pain after cesarean delivery using three simple questions. Anesthesiology. 2013 May;118(5):1170-9. doi: 10.1097/ALN.0b013e31828e156f. PMID 23485992
- [Derived] Street LM, Harris L, Curry RS, Eisenach JC. Capsaicin-induced pain and sensitisation in the postpartum period. Br J Anaesth. 2019 Jan;122(1):103-110. doi: 10.1016/j.bja.2018.09.026. Epub 2018 Nov 16. PMID 30579387